CLINICAL TRIAL: NCT06895954
Title: Shenzhen Hospital of Southern Medical University
Brief Title: The Clinical Study on Isoflavone Genistein in Restructuring the Gut Microbiota of Hyperlipidemia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Hospital of Southern Medical University (Other)
Responsible Party: Principal Investigator, Hongwei Zhou, Shenzhen Hospital of Southern Medical University, Shenzhen Hospital of Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NYSZYYEC2024K072R001
Record Dates: First submitted 2025-03-20; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-09

CONDITIONS: Hyperlipidemia
Keywords: Genistein; hyperlipidemia; gut microbiota; TMAO
MeSH Terms: conditions — Hyperlipidemias | interventions — Genistein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Genistein (Experimental): Dietary Supplement: Genistein Hyperlipidemia patients take a 125mg Genistein capsule daily, once a day.
  Interventions: Dietary Supplement: Genistein
- Control (No Intervention): The control group does not take the Genistein medication.

INTERVENTIONS:
Dietary Supplement: Genistein — Hyperlipidemia patients take a 125mg Genistein capsule daily, once a day.
  Arms: Genistein

SUMMARY:
: In preliminary animal experiments, we found that the soybean isoflavone compound Genistein could reduce serum TMAO levels in high-fat diet (HFD) mice, and this effect was dependent on the gut microbiota. Furthermore, we discovered that Genistein's regulatory effect on the gut microbiota in high-fat diet mice relies on the host colonic PKI-Nos2 pathway. Genistein is an isoflavone compound extracted from soybeans and is the most effective functional ingredient in soybean isoflavone products. It has multiple physiological functions, and several randomized controlled trials (RCTs) have shown that the intake of Genistein can effectively alleviate hyperlipidemia, obesity, metabolic syndrome, and cardiovascular diseases, suggesting its safety and efficacy as a clinical health supplement. Therefore, we aim to conduct clinical trials to further demonstrate that Genistein also influences the gut microbiota in hyperlipidemia patients, thereby reducing serum TMAO levels.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 30-65 years old, regardless of gender
* Abnormal donation and loan: including elevated total cholesterol and triglycerides, high triglycerides, and high triglycerides
* Volunteer to participate in clinical trials, understand and sign the informed consent form

Exclusion Criteria:

* Patients who do not meet the inclusion criteria
* Patients with gastrointestinal or chronic infectious diseases (i.e., diarrhea, Crohn's disease, ulcerative colitis, irritable bowel syndrome, diverticular disease, gastric or duodenal ulcer, hepatitis, HIV, cancer, etc.), or with a history of such diseases
* Chronic or acute kidney disease, eGFR < 50 in two or more laboratory tests in the past 6 months; diagnosis of cirrhosis or liver failure; hyperkalemia (defined as potassium > 5.4 in two or more laboratory tests in the past 6 months)
* Severe immunodeficiency (HIV positive, transplant patients, taking anti-rejection drugs, taking steroids for > 30 days, or receiving chemotherapy or radiotherapy in the past year)
* Alarm features such as weight loss, rectal bleeding, recent changes in bowel habits (< 3 months), or abdominal pain
* Patients with malignant diseases or any concomitant end-stage organ diseases
* Patients who have taken any antibiotics or dietary supplements (prebiotics, probiotics, fiber, resveratrol, fish oil, seed oil, ginkgo leaf, ginseng, fruit powder extract and DHA) within one month
* Patients who have taken any Chinese patent medicine or Chinese herbal decoction within one month
* Avoid eating seafood or fish 24 hours before each visit
* Vegetarian/vegan diet or food allergies or other food problems that will prevent the intake of research products
* Pregnant or preparing for pregnancy and breastfeeding women
* Allergic constitution, or known allergy to isoflavone genistein
* Participating in other drug clinical studies within 1 month
* According to the investigator's judgment, the patient cannot complete this study or cannot comply with the requirements of this study (due to management reasons or other reasons)

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-10-13 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Serum TMAO level | 12 months
Fecal TMA level | 12 months
Microbial flora structure | 12 months

SECONDARY OUTCOMES:
Serum CHOL level | 12 months
Serum TG level | 12 months
Serum LDLC level | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No